CLINICAL TRIAL: NCT03321656
Title: Impact of Envarsus XR® on Kidney Biopsy Subclinical Rejection and Blood Immunologic Profile
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Roberto Gedaly (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Roberto Gedaly, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42753
Record Dates: First submitted 2017-09-28; First posted 2017-10-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: * Treatment: Envarsus® 0.07-0.14 mg/kg/day every morning
  * Control: Generic tacrolimus 0.1-0.2 mg/kg/day in 2 divided doses given every 12 hours
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus (Active Comparator): 0.1 - 0.2 mg/kg/day in 2 divided doses every 12 hours orally
  Interventions: Drug: Tacrolimus
- Envarsus XR (Experimental): 0.07-0.14 mg/kg/day every morning orally
  Interventions: Drug: Envarsus XR

INTERVENTIONS:
Drug: Tacrolimus — 0.1-0.2 mg/kg/day orally divided into two doses every 12 hours orally
  Arms: Tacrolimus
Drug: Envarsus XR — 0.07-0.14 mg/kg/day every morning orally
  Arms: Envarsus XR

SUMMARY:
This will be a single center, prospective, open-label, randomized, controlled trial comparing Envarsus XR® to twice-daily tacrolimus. The targeted population will be patients with end stage renal disease listed for primary solitary kidney transplant. Transplant Surgery is not part of the study.

DETAILED DESCRIPTION:
Participants will be identified through the Department of Transplantation Surgery at the University of Kentucky. Participants will be pre-screened by the department for entry into the study. The investigator will determine if the participant meets study eligibility requirements.

The purpose of this research is to gather information on how safe and effective of Envarsus® is when compared to twice-daily tacrolimus. The results of this study will be shared with the company providing financial support for the study, the Food and Drug Administration and other federal agencies, if required.

All participants that successfully meeting inclusion criteria will be randomized (like the flipping of coin) to Envarsus vs. Tacrolimus at the time of transplant.

Participants will be randomized to one of two treatment arms. Treatment begins on post-op day 1.

* Treatment: Envarsus® 0.07-0.14 mg/kg/day every morning
* Control: Generic tacrolimus 0.1-0.2 mg/kg/day in 2 divided doses given every 12 hours

The total amount of time a person will be asked to volunteer for this study is 9-18 hours over the next 6 months.

Participants will need to complete 9 study visits each of these visits will take approximately 1-2 hours to complete. Participants will be given medication dosing diaries to complete throughout the study and will undergo 2 kidney biopsies.

Participants will be screened for HIV, Hepatitis B and Hepatitis C viruses.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English able to understand and provide informed consent.
* End stage renal disease listed for primary solitary kidney transplant.
* Willing to participate in the study and comply with study requirements as evidenced by signed IRB-approved informed consent.
* Female who are of childbearing potential will be asked to use 2 different medically acceptable methods of contraception for the duration of the study and at least 1 year post-infusion.

Exclusion Criteria:

* Previously undergone organ, tissue or cell transplant
* Allergic to Tacrolimus or MMF (Cellcept)
* Chronic use of blood thinners
* Previous chronic use of glucocorticoids or other immunosuppression, or biologic immunomodulators (prescribed for the treatment of serious inflammatory disorders)
* Significant or active infection
* Diagnosed with HIV, Hepatitis B or C, Herpes simplex virus, Varicella-Zoster virus, Epstein-Barr virus
* Have or have had cancer with in the past 3 years
* Have taken part in another study that involved an investigational drug within the last 12 months.
* Have a history of delayed or abnormal wound healing
* Are pregnant or breastfeeding
* Had a transfusion within the past 3 months
* Have or plan to be receive a live vaccination (intranasal influenza measles, mumps, rubella, oral polio, yellow fever, varicella)
* Are unable or unwilling to comply with study protocol or procedures.
* Current use anticoagulation medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
1. Change in the percentage of donor specific antibodies | Time of transplant and six months post-transplant
  We will check these donor specific antibodies to: HLA-A, -B and -C; or HLA-DR, -DQ and -DP. We will quantify the expression of these markers by Flow Cytometry analysis and reported as mean fluorescence intensity (MFI) units.
Changes in the percentage of blood immunologic markers | Time of transplant and six months post-transplant
  We will monitor the lymphocyte profile in blood in response to these 2 different treatments. The lymphocyte profile test will be performed by multi-parametric flow cytometry analysis with a panel of specific flourochrome-conjugated antibodies to selectively determine the following sub-populations:
  1. Circulating T cells: CD4/CD8 rates and determine the following CD4 subpopulations: effector TH1, TH2, TH9, Tfh, and regulatory/suppressor T cells.
  2. Circulating B cells (number and percentage of naïve, activated, memory and plasma B cells.
  3. Circulating NK cells (mature and immature)

SECONDARY OUTCOMES:
Changes in creatinine clearance | Time of transplant and six months post-transplant
  Baseline creatinine will be considered the creatinine plasma levels several days after transplantation once the kidney function is stabilized.

OTHER OUTCOMES:
Changes in GFR | 30 Days post transplant and months 3 and 6
  We will use the MDRD GFR equation to estimate glomerular filtration rate based on baseline creatinine and patient characteristics (age, gender and race)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Gedaly, MD, Principal Investigator — University of Kentucky
Locations (1):
- Deepa Valvi, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No